CLINICAL TRIAL: NCT04759898
Title: Direct Measurement of Motor Cortical Responses to Transcranial Direct Current Stimulation
Brief Title: Direct Measurement of Motor Cortical Responses to tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00073545
Record Dates: First submitted 2020-12-21; First posted 2021-02-18 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease; Chronic Stroke
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: In the first arm, Parkinson's disease and chronic stroke subjects will be investigated using noninvasive methods, including EEG and tDCS, respectively. In the second arm, a separate cohort of Parkinson's disease and chronic stroke subjects will be investigated using noninvasive methods, including EEG and sham tDCS, respectively. In the third arm, patients with Parkinson's disease will be investigated using electrocorticography (while undergoing surgery for deep brain stimulation) combined with tDCS.
Who Masked: Participant
Masking Description: In the first and second arms, prior to placement of electrodes, subjects will be randomized to either treatment or sham. This will occur using a random number generator with a binary choice determination (1 = stimulation; 2 = sham). Patients will be blinded to this choice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stimulation (noninvasive recording) (Active Comparator): Patients with Parkinson's disease or chronic stroke will be assigned to undergo EEG recording and transcranial direct current stimulation.
  Interventions: Device: transcranial direct current stimulation (noninvasive recording)
- Sham (noninvasive recording) (Sham Comparator): Patients with Parkinson's disease or chronic stroke will be assigned to undergo EEG recording and sham transcranial direct current stimulation.
  Interventions: Device: sham transcranial direct current stimulation (noninvasive recording)
- Stimulation (invasive recording) (Experimental): Patients with Parkinson's disease undergoing surgery for deep brain stimulation will be studied using electrocorticography combined with transcranial direct current stimulation
  Interventions: Device: transcranial direct current stimulation (invasive recording)

INTERVENTIONS:
Device: transcranial direct current stimulation (noninvasive recording) — Subjects will enter the EEG lab and be seated in a chair. The 26-electrode EEG array will be placed using a conductive paste. The electrodes will be connected to a clinical grade EEG machine used in standard of care routine EEG monitoring. Next, a soft cloth cap will be placed over the subject's head with the tDCS electrodes pre-positioned in place. The cap will be positioned so that the tDCS electrodes cover the scalp without disturbing the underlying EEG electrodes. Conducting gel will be applied in direct contact with the scalp to facilitate stimulation. In addition, lidocaine jelly will be added topically to provide local anesthesia. The tDCS electrodes will be connected to a low-current generator. Participants receive 2.0 milliamps in electrical stimulation from the tDCS machine for 20 minutes. The device will be manually controlled by study personnel assisting with the experiment. A virtual reality environment will be utilized to collect kinematic data during the study.
  Arms: Stimulation (noninvasive recording)
Device: sham transcranial direct current stimulation (noninvasive recording) — Subjects receiving sham undergo the same setup as the stimulation group with the exception that sham subjects experience stimulation for one minute only (30 second ramp-up to 2 milliamps immediately followed by 30 second ramp-down to 0 milliamps for the remaining 19 minutes). This provides similar sensory feedback to sham subjects that treatment subjects experience. The same electrode array, soft cloth cap, conducting gel application, and lidocaine are applied as in a stimulation subject. The tDCS electrodes will be connected to a low-current generator. A virtual reality environment will be utilized to collect kinematic data during the study.
  Arms: Sham (noninvasive recording)
Device: transcranial direct current stimulation (invasive recording) — Subjects are brought into the operating room. The scalp is prepped with a sterilizing solution. Following infiltration with local anesthetic and incision, a 6-contact electrocorticography strip is inserted into the burr hole covering primary motor cortex. Electrocorticography strip terminals are connected to an amplifier for signal recording. Gas-sterilized transcranial direct current stimulation electrodes are placed on the scalp directly overlying primary motor cortex. tDCS electrodes are connected to a low-current generator. During electrocorticographic recording, stimulation is turned on while subjects are asked to flex each arm. At the conclusion of the experiment, the electrocorticography strip and tDCS electrodes are removed and the surgery proceeds as planned.
  Arms: Stimulation (invasive recording)

SUMMARY:
Transcranial direct current stimulation (tDCS) has shown the potential to improve symptoms in patients with movement deficits, such as Parkinson's disease and chronic stroke. However, the effects of tDCS have so far not been proven on a wider scale due to lack of knowledge regarding exactly how tDCS works. This has limited the adoption of this potentially useful therapy for patients with Parkinson's disease, chronic stroke and other conditions affecting movement. The investigators hypothesize that by studying the effects of tDCS in subjects performing a motor task, the brain signals mediating improvements in motor control will be identified. The investigators will use both noninvasive and invasive methods to explore this hypothesis. The investigators expect this combined approach to broaden understanding of tDCS application in conditions affecting movement and possibly lead to therapeutic advances in these populations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Previous consent to be contacted regarding potential participation in a research study at Medical University of South Carolina

Exclusion Criteria:

* Subjects unable to actively participate in the consent process physically and/or cognitively
* Pregnancy
* Presence of scalp injury or disease
* Prior history of seizures
* Metal implants in head or neck
* Prior intracranial surgery
* Prior brain radiotherapy
* Prior history of intracranial tumor, intracranial infection or cerebrovascular malformation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in primary motor cortical (PriMC) beta oscillations during cued arm reaching in relation to anodal tDCS activation | Subjects will undergo baseline EEG recording 5 min before tDCS starts, during tDCS (5 min after stimulation starts) and 5 min after tDCS stimulation ends. Measurements will be made similarly during sham stimulation.
  EEG is used to track beta spectral power during a cued motor task in conjuction with transcranial direct current stimulation or sham
Change in primary motor cortical (PriMC) beta oscillations during arm flexion in relation to anodal tDCS activation | Subjects will undergo baseline ECoG recording 5 min before tDCS starts, during tDCS (5 min after stimulation starts) and 5 min after tDCS stimulation ends. Measurements will be made similarly during sham stimulation.
  ECoG is used to track beta spectral power during an arm flexion task in conjuction with transcranial direct current stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Nathan C Rowland, MD,PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No